CLINICAL TRIAL: NCT04146792
Title: Expand Your Horizon: An Online Writing Intervention for Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Society for the Psychological Study of Social Issues (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20016491
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Body Image

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- body acceptance program (Experimental)
  Interventions: Behavioral: body acceptance program
- writing creativity program (Active Comparator)
  Interventions: Behavioral: writing creatively program

INTERVENTIONS:
Behavioral: body acceptance program — Complete 3 writing exercises over the course of week. Each writing exercise will take approximately 15 minutes to complete
  Arms: body acceptance program
Behavioral: writing creatively program — Complete 3 writing exercises over the course of week. Each writing exercise will take approximately 15 minutes to complete
  Arms: writing creativity program

SUMMARY:
The purpose of this research study is to test a new writing-based intervention that helps young adult women increase their body acceptance and fosters creativity.

DETAILED DESCRIPTION:
In this study, participants will be asked to do the following things:

1. Complete 3 writing exercises over the course of week. Each writing exercise will take approximately 15 minutes to complete
2. ~1-hour long online surveys immediately after the program (1 week), and 1 week after the program. Questions will ask about eating behaviors and attitudes, body image, feelings of weight stigma, and mental health.
3. Be contacted through email to remind participants to complete the writing assignments/survey

ELIGIBILITY:
Inclusion Criteria:

* women ages 18 to 25 years
* enrolled in postsecondary education at VCU
* endorse some degree of WBI (as measured by the WBI-M) or body image concerns

Exclusion Criteria:

* men
* pregnant women

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Change in weight bias internalization (WBI) | baseline to 2 weeks
  The Modified Weight Bias Internalization Scale (WBIS-M) is a modified version of the Weight Bias Internalization Scale that was adapted for use with individuals across the weight spectrum. The WBIS-M measures the degree to which individuals apply weight-based stereotypes to themselves and use those to guide their weight self-evaluations. Items are rated on a 7-point scale, with higher scores reflecting greater degrees of weight bias internalization.

SECONDARY OUTCOMES:
Change in body functionality appreciation | baseline to 2 weeks
  Body functionality appreciation will be assessed using the Functionality Appreciation Scale (FAS). The Functionality Appreciation Scale (FAS) is a 7-item scale that measures appreciation for the functionality of one's body, which is believed to help offset appearance concerns. Items are rated on a 5-point scale with higher scores reflecting greater appreciation for the functionality of one's body.
Change in body image dissatisfaction | Baseline to 2 weeks
  Body dissatisfaction will be measured using Body-Image Ideals Questionnaire (BIQ. The BIQ is a 22-item measure that assesses appearance satisfaction. This scale examines both perceived discrepancy between one's body image ideal and current appearance as well as the importance of appearance to one's self-concept.
Change in objectified body consciousness | Baseline to 2 weeks
  Objectified body consciousness will be assessed using the Body Consciousness Scale (OBCS). This is a 24-item measure that assesses the degree to which one experiences their body as an object.
Change in self-compassion | Baseline to 2 weeks
  Self-Compassion will be assessed using the Self-Compassion Scale-Short Form (SCS-SF). This is a 12-item measure that assesses the degree to which one is able to hold her or his own feelings of suffering with a sense of warmth, connection, and concern
Change in depression | Baseline to 2 weeks
  Depression will be assessed using the depression subscale of the Depression, Anxiety, and Stress Scales (DASS-21). This measure asks participants to rate the frequency and severity of negative emotions over the previous week. Items are rated on a four-point scale (0 = did not apply to me at all, 3 = applied to me very much or most of the time).
Change in anxiety | Baseline to 2 weeks
  Anxiety will be assessed using the anxiety subscale of the Depression, Anxiety, and Stress Scales (DASS-21). This measure asks participants to rate the frequency and severity of negative emotions over the previous week. Items are rated on a four-point scale (0 = did not apply to me at all, 3 = applied to me very much or most of the time).
Change in stress | Baseline to 2 weeks
  Stress will be assessed using the stress subscale of the Depression, Anxiety, and Stress Scales (DASS-21). This measure asks participants to rate the frequency and severity of negative emotions over the previous week. Items are rated on a four-point scale (0 = did not apply to me at all, 3 = applied to me very much or most of the time).
Change in healthcare stress | Baseline to 2 weeks
  Healthcare Stress will be assessed using a scale created by weight stigma researchers. This is a five-item scale that was originally adapted for a study on healthcare anxiety in higher weight women. Participants use a 10-point scale (1 = No stress, 10 = Very stressed) to indicate their level of stress when thinking about numerous healthcare encounters.
Change in healthcare avoidance | Baseline to 2 weeks
  Healthcare Avoidance will be assessed by a four-item scale that measures how often someone avoids healthcare. The measure was adapted for the current study such that we deleted an item about mammograms because it is not relevant to this age group. Also, given the short follow-up period, we assumed that participants' healthcare utilization would not change over the course of the study. Thus, we also modified the rating scale to reflect intent to avoid healthcare. Participants will use a five-point scale (1 = Extremely Likely, 5 = Extremely Unlikely) to indicate their likelihood to utilize numerous healthcare encounters.
Change in physical activity acceptance | Baseline to 2 weeks
  Physical activity acceptance will be assessed using the Physical Activity Acceptance Questionnaire (PAAQ). The PAAQ is a 10-item measure that assesses participants' ability to accept the discomfort associated with exercising.
Change in global eating disorder symptoms | Baseline to 2 weeks
  Disordered eating will be assessed using the Eating Disorder Examination - Questionnaire (EDE-Q). The EDE-Q is a 28-item self-report version of the Eating Disorder Examination that measures frequency of disordered eating cognitions and behaviors experienced in the previous 28 days. Participants rate the number of days behaviors have occurred in the last 28 days, with 0 = no days and 6 = every day. Yes/no questions identify the presence of compensatory and binge behaviors and participants indicate the frequency of these behaviors over the last 28 days. Higher EDE-Q scores indicate greater eating pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Mazzeo, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Individual level data will not be shared other researchers. Access to all data will be limited to study personnel.